CLINICAL TRIAL: NCT01566201
Title: The Effect of Inhibition of Interleukin-1 Activity on Vascular and Left Ventricular Function in Patients With Coronary Artery Disease and Coexistent Rheumatoid Arthritis
Brief Title: Effects of Interleukin-1 Inhibition on Vascular and Left Ventricular Function in Rheumatoid Arthritis Patients With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Assistant Professor in Cardiology, University of Athens
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RCT-RACAD-ATTIKON-01
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Rheumatoid Arthritis; Coronary Artery Disease; Inflammation
Keywords: Arterial stiffness; Endothelial function; Left ventricular function; Apoptosis; Nitrooxidative stress
MeSH Terms: conditions — Arthritis, Rheumatoid; Coronary Artery Disease; Inflammation | interventions — Interleukin 1 Receptor Antagonist Protein; Water; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- anakinra (Active Comparator)
  Interventions: Drug: anakinra
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: anakinra — Inhibition of Interleukin-1 activity by anakinra (Kineret®) 100mg od, sc injection
  Other Names: Kineret® (anakinra)
  Arms: anakinra
Drug: placebo — water for injection
  Other Names: water for injection
  Arms: placebo

SUMMARY:
Inhibition of interleukin-1 (IL-1) activity in patients with RA without CAD ameliorates vascular and LV function. Moreover, data from species shows beneficial effect of this treatment on LV function after experimental myocardial infarction. The purpose of this study is to investigate whether anakinra, an IL-1 receptor antagonist, improves vascular and left ventricular (LV) function in patients with coronary artery disease (CAD) and coexistent rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
The inflammatory processes observed in patients with rheumatoid arthritis (RA) are strongly linked to enhanced interleukin-1 (IL-1) activity. Increased IL-1 activity causes myocardial cell damage and endothelial dysfunction. The adverse effects of IL-1 on myocardial and endothelial cells are mediated by an enhanced nitrooxidative stress and the promotion of apoptotic cardiomyocyte death through increased nitrooxidative stress and inflammation. Anakinra, a recombinant form of human IL-1 receptor antagonist, is commonly used for the treatment of RA. Experimental data indicates that administration of anakinra after acute myocardial infarction ameliorates cardiac remodeling by reducing cardiomyocyte apoptosis. Moreover, in our previous studies we have shown that treatment with anakinra reduces IL-1-mediated nitrooxidative stress and apoptotic markers leading to an improvement in Tissue Doppler and speckle tracking-derived parameters of left ventricular (LV) function in RA patients. However it has not been defined whether inhibition of IL-1 activity by anakinra shows beneficial effects on endothelial, coronary, arterial and LV systolic and diastolic function in patients with coronary artery disease (CAD).

For this purpose, we studied 60 patients with CAD and coexistent RA (American Rheumatism Association criteria) as well as 20 patients with RA and without CAD. All the above subjects had an inadequate response to disease modifying antirheumatic drugs (DMARDs) and corticosteroids and were going to initiate treatment with IL-1 activity inhibitor (anakinra). All patients were on treatment with statins and cardioactive medications respectively, for the last 6 months. In the 20 patients with only RA, the presence of CAD was excluded with a non-invasive test and/or a negative recent coronary arteriogram.

In a double-blind, placebo-controlled fashion, all patients were randomized to receive a single injection of anakinra(100 mg s.c.) or placebo. After 48-hours patients were crossed over to the alternate treatment (placebo or anakinra) and measurement of the examined markers was repeated. The 48h interval between the 2 consecutive studies was decided to secure a sufficient wash-out period of anakinra in accordance to the drug's half-life time.

Twenty asymptomatic subjects matched for age and sex as the RA patients and with a normal ECG, echocardiogram, and treadmill test were selected as healthy control subjects among subjects attending the cardiology outpatients' clinic.

At baseline in all RA subjects and controls as well as 3-hours after the single injection of anakinra in RA subjects, we assessed by means of echocardiography the following parameters a) the LV dimensions,fractional shortening and wall motion score index (WMSI) b) the systolic (Sm), early diastolic (Em) and late diastolic (Am) myocardial velocities of the mitral annulus by using of tissue Doppler (TDI) as well as the ratio of E wave of the mitral inflow measured by pulsed wave Doppler to the mean Em as an index of LV diastolic filling pressures c) the LV longitudinal, circumferential and radial strain and strain rate, as well as Global Longitudinal strain and Torsion using speckle tracking echocardiography d) the coronary flow reserve (CFR)after adenosine infusion to assess coronary vasomotor function e) the flow-mediated endothelial-dependent dilation of the brachial artery (FMD) to assess peripheral endothelial function f) the diameters of aorta at systole and diastole to calculate the aortic strain as an index of local aortic properties. At the same time periods, we measured in blood samples a) nitrotyrosine (NT), protein carbonyls (PC)and malondialdehyde(MDA)to assess nitrooxidative stress b)soluble Fas and Fas-ligand )to assess apoptosis c) interleukin-1b and tumor necrosis factor-a to assess inflammation

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis and coexistent coronary artery disease or without CAD who had an inadequate response to disease modifying antirheumatic drugs (DMARDs) and corticosteroids and were going to initiate treatment with interleukin-1 inhibitor.

Exclusion Criteria:

* Familiar hyperlipidemia
* Diabetes mellitus
* Chronic obstructive pulmonary disease or asthma, moderate or severe valvular heart disease, primary cardiomyopathies,malignant tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Improvement in vascular and left ventricular function after anakinra | 3 hours after treatment
  Improvement in vascular and left ventricular function after administration of anakinra compared to placebo

SECONDARY OUTCOMES:
Reduction of nitrooxidative stress and apoptosis after anakinra treatment | 3 hours after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; Stavros Tzortzis, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; John P. Lekakis, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; Ioanna Andreadou, Dr, Principal Investigator — Department of Pharmaceutical Chemistry, University of Athens Medical School, Greece; Ioannis Paraskevaidis, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece; Maria Anastasiou-Nana, MD, Principal Investigator — 2nd Cardiology Department, University of Athens, Greece
Locations (1):
- "Attikon" University General Hospital, Haidari, Athens, Attica, Greece

REFERENCES:
- [Derived] Ikonomidis I, Tzortzis S, Andreadou I, Paraskevaidis I, Katseli C, Katsimbri P, Pavlidis G, Parissis J, Kremastinos D, Anastasiou-Nana M, Lekakis J. Increased benefit of interleukin-1 inhibition on vascular function, myocardial deformation, and twisting in patients with coronary artery disease and coexisting rheumatoid arthritis. Circ Cardiovasc Imaging. 2014 Jul;7(4):619-28. doi: 10.1161/CIRCIMAGING.113.001193. Epub 2014 Apr 29. PMID 24782115